CLINICAL TRIAL: NCT05904366
Title: Magnetic Resonance Spectroscopy in Acid Sphingomyelinase Deficiency
Acronym: MONACO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eline C. B. Eskes (Other)
Responsible Party: Sponsor-Investigator, Eline C. B. Eskes, MD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022.0444
Record Dates: First submitted 2023-06-06; First posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Asmd, Visceral Type
MeSH Terms: conditions — Niemann-Pick Disease, Type B

STUDY DESIGN:
Intervention Model Description: Cross-sectional pilot study in which MRS and MRE measurements of ASMD patients will be compared to measurements in healthy subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients (Other): Participants will undergo an MRI with MR Spectroscopy (MRS) and MR Elastography (MRE) measurements
  Interventions: Diagnostic Test: MR Spectroscopy (MRS); Diagnostic Test: MR Elastography (MRE)
- Healthy controls (Other): Participants will undergo an MRI with MR Spectroscopy (MRS) and MR Elastography (MRE) measurements
  Interventions: Diagnostic Test: MR Spectroscopy (MRS); Diagnostic Test: MR Elastography (MRE)

INTERVENTIONS:
Diagnostic Test: MR Spectroscopy (MRS) — MR Spectroscopy (MRS)
Diagnostic Test: MR Elastography (MRE) — MR Elastography (MRE) with a device that induces shear waves in the body. This device is placed upon the abdomen of the subject and is hold in place by straps. The device will produce low-frequency vibrations (e.g. 30-60 Hz) which are not painful to the participant. A declaration of conformity and a safety document are provided in the study dossier.

SUMMARY:
The goal of this study is to assess the ability of MRI techniques to detect early stages of lipid accumulation in the liver of ASMD patients with the chronic visceral subtype compared to healthy subjects.

Participants will undergo an MRI with MR Spectroscopy (MRS) to measure lipid accumulation (steatosis) and MR Elastography (MRE) to measure liver stiffness (fibrosis).

DETAILED DESCRIPTION:
Rationale: Acid sphingomyelinase deficiency (ASMD) is a rare lysosomal storage disorder caused by a deficiency of sphingomyelinase resulting in accumulation of the sphingolipid sphingomyelin (SM) in the liver, spleen and lungs. Accumulation of SM in the liver leads to liver fibrosis in a subset of ASMD patients. Enzyme replacement therapy (ERT, olipudase alfa, Sanofi Genzyme) is currently investigated in a phase 2/3 trial and recently received market authorization by the EMA and FDA. As ASMD is a slowly progressive disease, detection of early stages of SM storage in the liver might aid in identifying patients at risk for major complications who would benefit from therapy. Two magnetic resonance (MR) based techniques might be of interest: MR Spectroscopy (MRS) to measure lipid accumulation (steatosis) and MR Elastography (MRE) to measure liver stiffness (fibrosis).

Objective: To assess the ability of MRI techniques to detect early stages of lipid accumulation in the liver of ASMD patients with the chronic visceral subtype compared to healthy subjects.

Study design: Cross-sectional pilot study in which MRS and MRE measurements of ASMD patients will be compared to measurements in healthy subjects. All ASMD patients who participate will undergo an MRI during their yearly assessments. Patients eligible for therapy will also undergo an MRI after one year of treatment.

Study population: All adult patients with ASMD visiting the outpatient clinic for metabolic disorders of the Amsterdam UMC will be invited to participate. Participating ASMD patients will be matched to healthy controls based on age, sex and BMI in a ratio of 1:1.

Main study endpoint: Fat fraction in volume percentage (%) of liver tissue of ASMD patients measured with MRS compared to values of healthy subjects.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The MRI procedure yields no risk: at most patients might feel uncomfortable lying in the tight space. Patients and healthy subjects will not directly benefit from participation in the study. The results of the study may improve clinical care in the future.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* The patient has biochemically proven ASMD (preferably genetically confirmed)
* The patient is willing and able to provide written informed consent prior to the study-related procedure.
* The patient is ≥ 18 years of age

Healthy controls:

* The individual is willing and able to provide written informed consent prior to the study-related procedure
* The individual is ≥ 18 years of age
* General good health as determined by medical history

Exclusion Criteria:

Patients and healthy controls:

* Inability to adhere to the study protocol
* Inability to undergo an MRI procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2023-05-05 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Fat fraction in volume percentage measured with MRS-PDFF | 1 year
  Fat fraction in volume percentage measured with MRS-PDFF of ASMD patients compared to age-, sex, and BMI-matched healthy subjects.

SECONDARY OUTCOMES:
Liver stiffness in kPa measured with MRE | 1 year
  Liver stiffness in kPa measured with MRE of ASMD patients compared to age-, sex, and BMI-matched healthy subjects.
Correlations between fat fraction and/or liver stiffness and liver parameters | 1 year
  Correlations between fat fraction and/or liver stiffness and liver parameters (i.e. liver stiffness measured with fibroscan, liver volume and plasma ALT and AST levels)
Correlations between fat fraction and/or liver stiffness and general disease parameters | 1 year
  Correlations between fat fraction and/or liver stiffness and general disease parameters (i.e. spleen volume, CO diffusion capacity, plasma LSM, LSM-509 and chitotriosidase levels)

CONTACTS AND LOCATIONS:
Overall Officials: Carla EM Hollak, prof dr, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); xx xx xx, xx, Study Director
Locations (1):
- Amsterdam UMC, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Research data will be submitted as articles to peer-reviewed journals. Also, an abstract of our research data reporting our findings will be submitted for presentations on scientific, public and/or patient organization meetings for (oral) presentation(s).